CLINICAL TRIAL: NCT01663259
Title: Reduced-intensity Therapy for Advanced Oropharyngeal Cancer in Non-smoking Human Papilloma Virus (HPV)-16 Positive Patients
Brief Title: Reduced-intensity Therapy for Oropharyngeal Cancer in Non-smoking HPV-16 Positive Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan Rogel Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UMCC 2009.078; HUM00032219 (Other: University of Michigan IRBMED); NCT01649414 (obsolete NCT alias)
Record Dates: First submitted 2012-07-23; First posted 2012-08-13 (Estimated); Results first posted 2020-10-26 (Actual); Last update posted 2021-01-19 (Actual); Status verified 2020-12

CONDITIONS: Squamous Cell Carcinoma of the Oropharynx; HPV
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — Cetuximab; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Cetuximab (Experimental)
  Interventions: Drug: Cetuximab; Radiation: Radiotherapy

INTERVENTIONS:
Drug: Cetuximab — Before Radiotherapy patients you will receive a single loading dose of cetuximab. Patients will also have two additional biopsies before and after cetuximab to determine how the tumor is affected. A Cetuximab infusion will also be delivered once a week during radiotherapy.Radiation will be started (70 Gy in 35 fractions over 7 weeks to the gross tumor, 50-60 Gy to subclinical target volumes) five days a week until the total dose of radiation prescribed by the doctor is reached. Radiation will be delivered concurrent with weekly cetuximab 250 mg/m2, delivered on Monday or Tuesday each week. In order to evaluate swallowing problems from radiotherapy, patients will undergo an evaluation of swallowing by videofluoroscopy (VF). Quality of Life questionnaires will be given before therapy and periodically up to 36 months after therapy. In order to assess if the tumor was completely eradicated, CT-PET scan will be performed 3 months after the completion of therapy.
Radiation: Radiotherapy — Radiation will be started (70 Gy in 35 fractions over 7 weeks to the gross tumor, 50-60 Gy to subclinical target volumes) five days a week until the total dose of radiation prescribed by the doctor is reached. Radiation will be delivered concurrent with weekly cetuximab 250 mg/m2, delivered on Monday or Tuesday each week.

SUMMARY:
Taking into account the excellent prognosis of patients with HPV-positive oropharyngeal cancer with < 10 pack-year smoking, the investigators hypothesize that reducing the intensity of therapy for these patients will reduce treatment sequelae, notably long-term dysphagia, without affecting their cure rates. The main Aim is to assess whether reducing treatment intensity, by replacing concurrent chemotherapy with cetuximab, will indeed achieve improved long-term toxicity.

The primary objectives include the following: to confirm that reducing treatment intensity in patients with HPV-related oropharyngeal cancer and < 10 pack-year smoking history by replacing concurrent chemotherapy with concurrent cetuximab, does not significantly increase the proportion of patients whose tumors recur, compared to our previous experience in similar patients receiving chemo-RT and to compare the toxicity in patients receiving cetuximab-RT to similar patients treated with 7 weeks of chemotherapy concurrent with RT ("standard therapy") in UMCC 2-21.

DETAILED DESCRIPTION:
The investigators have shown in past experience a high success in getting rid of oropharyngeal cancer (tonsil or base of tongue cancer) using chemotherapy and radiation therapy in patients who have not smoked, or only smoked a minimal amount of cigarettes or equivalent. In these patients, the cancer is thought to be caused by a virus (Human Papilloma Virus, or HPV). HPV is a virus that infects the epidermis (outermost layer of skin) and mucous membranes of humans. In general, patients with HPV-related cancer such as yours have a better prognosis compared with patients whose tumors are smoking-related. Taking into account the good prognosis, it is possible that reducing the intensity of therapy will not affect the high rate of tumor control, while reducing the side-effects of therapy. In this study, the investigators plan to reduce the intensity of treatment by replacing the currently used chemotherapy drugs with an FDA approved drug, cetuximab, which is a monoclonal antibody to a growth factor which helps cancer cells grow. By opposing the effect of the growth factor, cetuximab may help radiotherapy kill cancer cells without a lot of effect on the normal tissue. It differs from chemotherapy in its more selective activity against tumors compared to normal tissue Cetuximab has the chance to preserve the high rate of success in killing the tumor but may reduce the side effects and complications of therapy in comparison to chemotherapy drugs.

The investigators would also like to know if taking cetuximab has any effect on certain cancer-related molecules in the cancer and the normal cells inside the cheek. They would like to test this by taking a small biopsy of the tumor, as well as a swab of the inside of the cheek, before and shortly after the start of therapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have pathologically-confirmed, previously untreated,stage III-IV(excluding N3 or T4) squamous cell carcinoma of the oropharynx, without evidence of distant metastasis
* Pretreatment tumor biopsy with sufficient tumor for HPV or p16 analysis is required. The tumor must be HPV(+) or p16(+)

Smoking history <10 pack-year or equivalent (including cigarettes, cigars, pipes, chewing tobacco, and/or marijuana). One cannabis joint is equivalent to 5 cigarettes. (Aldington etal, Thorax 2007; 62:1058-1063). Smoking status definitions (National Health Interview Survey and Behavioral Risk Factor Surveillance System (Nelson DE etal al, Am J Pub Health 2003;93:1335):

* Smokers: smoking now every day or some days in past month
* Quitters: at least 100 cigarettes/lifetime and not smoking in the past 1-12 months
* Former smoker: at least 100 cigarettes/lifetime and not smoking >12 months
* Never smokers: <100 cigarettes (or equivalent)/lifetime

  * KPS > 80 (see Appendix A)
  * Patients must undergo pre-treatment endoscopic tumor staging and PET-CT scanning
  * Laboratory criteria:
* WBC > 3500/ul
* granulocyte > 1500/ul
* Platelet count > 100,000/ul
* Total Bilirubin < 1.5 X ULN
* AST and ALT < 2.5 X ULN

  * Creatinine clearance >30 cc/min
  * Patients must sign study specific informed consent
  * Patients must have, in the opinion of a treating physician, tumor that is accessible to biopsy in the clinic.

Exclusion Criteria:

* Prior head and neck malignancy or history of other prior non-head and neck malignancy (excluding skin cancer and early stage treated prostate cancer) within the past 3 years
* Prior head and neck radiation or chemotherapy
* Any medical or psychiatric illness, which in the opinion of the principal investigator, would compromise the patient's ability to tolerate this treatment or limit compliance with study requirements
* Patients residing in prison
* Patients with prior anti-epidermal growth-factor receptor antibody therapy (antibody or small molecule)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2011-01 (Actual); Primary Completion 2019-09 (Actual); Study Completion 2019-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michelle Mierzwa, MD, Principal Investigator — University of Michigan Rogel Cancer Center
Locations (1):
- Radiation Oncology , University of Michigan Health System, Ann Arbor, Michigan, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 43 patients consented, but one never began treatment.
Groups:
- Cetuximab + Radiotherapy: Patients received a single loading dose public) of cetuximab 400 mg/m (Day 0), then weekly cetuximab 250 mg/m concurrent with radiation. Within approximately 4 days after first (loading) dose of cetuximab, patients received radiation administered as 70 Gy in 35 fractions to the gross tumor, 50-60 Gy to subclinical target volumes.
Period: Overall Study
Arm/Group | Cetuximab + Radiotherapy
Started | 42
Completed | 42
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Cetuximab + Radiotherapy
Number analyzed (Participants) | 42
Age, Continuous [Mean (Full Range); unit: years] | 58 [48 to 76]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 36
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 40
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 41
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 42
Smoking [Count of Participants; unit: Participants]
  Yes, current | 1
  Yes, past | 5
  No | 36
Cancer Location [Count of Participants; unit: Participants]
  Oropharynx | 42
  Oral Cavity | 0
  Auditory Canal | 0
  Hypopharynx | 0
  Unknown Primary | 0
HPV Status [Count of Participants; unit: Participants]
  Positive | 42
  Negative | 0

OUTCOME MEASURES:

1. Primary Outcome: Rate of Recurrence
Description: Number of patients whose tumors recur (includes local, regional, and distant recurrence; and second primaries).
  Note: Research indicates that freedom from local and regional progression (FFLRP) is a more meaningful measure. Therefore, the percentage of patients with FFLRP is included below as a Post-Hoc measure.
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Groups:
- Cetuximab + Radiotherapy: Patients received a single loading dose of cetuximab and a Cetuximab infusion delivered once a week during radiotherapy.
Arm/Group | Cetuximab + Radiotherapy
Number analyzed (Participants) | 42
Participants | 8

2. Secondary Outcome: Number of Participants With Adverse Events
Description: In order to evaluate the toxicity in patients receiving cetuximab-RT, adverse events were clustered into three categories: None, Mild-Moderate (grade 1 or 2), and Severe (grade 3 or 4). Graded according to the Common Terminology Criteria for Adverse Events version 4.0 (CTCAE v4).
Time Frame: 3 years
Measure: Count of Participants; unit: Participants
Arm/Group | Cetuximab + Radiotherapy
Number analyzed (Participants) | 42
Participants
  None | 0
  Mild-Moderate | 14
  Severe | 28

3. Secondary Outcome: Treatment Related Toxicities
Description: Toxicities are measured by number of participants who experience one or more types or indicator of toxicity, shown as all grades and grades 3-4. As each participant could have multiple toxicities, the number of incidents outnumbers the number of participants. Toxicities graded according to the CTCAE v4.
Time Frame: 3 years
Measure: Number; unit: participants
Arm/Group | Cetuximab + Radiotherapy
Number analyzed (Participants) | 42
participants
  All Grades : Cutaneous Toxicity | 38
  All Grades : Mucositis | 42
  All Grades : Dysphagia | 37
  All Grades : Hematologic Toxicity | 13
  Grades 3-4 : Cutaneous Toxicity | 3
  Grades 3-4 : Mucositis | 19
  Grades 3-4 : Dysphagia | 7
  Grades 3-4 : Hematologic Toxicity | 6

4. Secondary Outcome: Mean Change in Tumor Epidermal Growth Factor Receptor (EGFR)
Description: The ratio (fold change) of tumor EGFR post/pre loading dose of cetuximab. Reported as the mean of fold changes across all participants who had an evaluable tumor sample.
Time Frame: Day 7
Population: 8 participants had a sample size sufficient for EGFR analysis.
Measure: Mean (Full Range); unit: fold change
Arm/Group | Cetuximab + Radiotherapy
Number analyzed (Participants) | 8
fold change | 1.2 [0.1 to 2.5]

5. Secondary Outcome: Mean Change in Tumor Phosphorylated EGFR (pEGFR)
Description: The ratio (fold change) of tumor pEGFR post/pre loading dose of cetuximab. Reported as the mean of fold changes across all participants who had an evaluable tumor sample.
Time Frame: Day 7
Population: 2 participants had a sample size sufficient for pEGFR analysis.
Measure: Mean (Full Range); unit: fold change
Arm/Group | Cetuximab + Radiotherapy
Number analyzed (Participants) | 2
fold change | 0.55 [0.5 to 0.6]

6. Secondary Outcome: Change in Tumor EGFR Level Relative to EGFR in Normal Mucosa
Description: Normal mucosa EGFR was assessed for comparison with EGFR in tumor sample. The fold change in tumor EGFR level post/pre loading dose of cetuximab, relative to fold change in normal mucosa EGFR level post/pre loading dose of cetuximab was summarized across all participants who had an evaluable tumor sample and normal mucosa sample. The value reported is the ratio of fold change in tumor/fold change in buccal EGFR.
Time Frame: Day 7
Population: 7 participants had a sample size sufficient for EGFR analysis.
Measure: Mean (Full Range); unit: ratio
Arm/Group | Cetuximab + Radiotherapy
Number analyzed (Participants) | 7
ratio | 1.31 [0.1 to 2.5]

7. Post Hoc Outcome: Disease Free Survival Rate
Description: Percentage of participants who survived without recurrent disease, from the time of enrollment to 1 and 2 years.
Time Frame: 2 years
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Cetuximab + Radiotherapy
Number analyzed (Participants) | 42
Percentage of participants
  1 year | 85.7 [75.8 to 97]
  2 year | 81 [69.9 to 93.7]
Statistical Analysis 1: Comparison: Cetuximab + Radiotherapy; Test type: Other; Estimates of proportion event-free at 1 and 2 years calculated using Kaplan-Meier methods, and the 2-sided, 95% confidence intervals were calculated by the Greenwood method. All analyses were performed using SAS v9.4 software and R version 3.5.2

8. Post Hoc Outcome: Overall Survival Rate
Description: Percentage of participants alive at 1 and 2 years after enrollment.
Time Frame: 2 years
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Cetuximab + Radiotherapy
Number analyzed (Participants) | 42
Percentage of participants
  1 year | 97.6 [93.1 to 100]
  2 year | 95.2 [89 to 100]
Statistical Analysis 1: Comparison: Cetuximab + Radiotherapy; Test type: Other; Survival proportion estimates at 1 and 2 years were calculated using Kaplan-Meier methods, and the 2-sided, 95% confidence intervals calculated by the Greenwood method. All analyses were performed using SAS v9.4 software and R version 3.5.2

9. Post Hoc Outcome: Freedom From Local Regional Progression (FFLRP)
Description: Percentage of participants without first local or regional recurrence at one and at two years from the time of enrollment. Local recurrence refers to mouth or throat; regional recurrence refers to nearby lymph nodes.
Time Frame: 2 years
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cetuximab + Radiotherapy
Number analyzed (Participants) | 42
percentage of participants
  1 year | 87.9 [75.8 to 97]
  2 years | 87.9 [69.9 to 93.7]
Statistical Analysis 1: Comparison: Cetuximab + Radiotherapy; Test type: Other; Estimates of proportion LRP event-free at 1 and 2 years were calculated using Kaplan-Meier methods, and the 2-sided, 95% confidence intervals calculated by the Greenwood method. All analyses were performed using SAS v9.4 software and R version 3.5.2

ADVERSE EVENTS:
Time Frame: 3 years
Groups:
- Cetuximab: Patients received a single loading dose of cetuximab and a Cetuximab infusion delivered once a week during radiotherapy.
Arm/Group | Cetuximab
All-Cause Mortality (participants affected / at risk) | 2/42
Serious Adverse Events (participants affected / at risk) | 9/42
Other Adverse Events (participants affected / at risk) | 42/42
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cetuximab (N=42)
Colitis (Gastrointestinal disorders) | 1 (1)
Gastrointestinal disorders - other (Gastrointestinal disorders) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 4 (4)
Nausea (Gastrointestinal disorders) | 1 (1)
Oral pain (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Lung infection (Infections and infestations) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 1 (1)
Lymphocyte count decreased (Investigations) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Cognitive disturbance (Nervous system disorders) | 1 (1)
Confusion (Psychiatric disorders) | 1 (1)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cetuximab (N=42)
Anemia (Blood and lymphatic system disorders) | 5 (5)
Lymph node pain (Blood and lymphatic system disorders) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 3 (5)
External ear inflammation (Ear and labyrinth disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 9 (9)
Diarrhea (Gastrointestinal disorders) | 4 (6)
Dry mouth (Gastrointestinal disorders) | 40 (92)
Dyspepsia (Gastrointestinal disorders) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 40 (96)
Esophagitis (Gastrointestinal disorders) | 41 (84)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 2 (2)
Gastrointestinal disorders - Other (Gastrointestinal disorders) | 21 (51)
Mucositis oral (Gastrointestinal disorders) | 42 (115)
Nausea (Gastrointestinal disorders) | 24 (46)
Oral pain (Gastrointestinal disorders) | 6 (15)
Salivary duct inflammation (Gastrointestinal disorders) | 12 (18)
Vomiting (Gastrointestinal disorders) | 9 (16)
Chills (General disorders) | 6 (7)
Facial pain (General disorders) | 1 (1)
Fatigue (General disorders) | 26 (45)
Fever (General disorders) | 4 (5)
Flu like symptoms (General disorders) | 1 (1)
Infusion related reaction (General disorders) | 3 (3)
Pain (General disorders) | 1 (1)
Allergic reaction (Immune system disorders) | 1 (1)
Lung infection (Infections and infestations) | 1 (1)
Papulopustular rash (Infections and infestations) | 2 (4)
Paronychia (Infections and infestations) | 3 (3)
Dermatitis radiation (Injury, poisoning and procedural complications) | 38 (64)
Fall (Injury, poisoning and procedural complications) | 1 (1)
Alanine aminotransferase increased (Investigations) | 9 (13)
Alkaline phosphatase increased (Investigations) | 2 (2)
Aspartate aminotransferase increased (Investigations) | 7 (9)
Blood bilirubin increased (Investigations) | 3 (3)
Creatinine increased (Investigations) | 1 (1)
Lymphocyte count decreased (Investigations) | 14 (43)
Platelet count decreased (Investigations) | 4 (4)
Urine output decreased (Investigations) | 2 (2)
Weight loss (Investigations) | 11 (14)
White blood cell decreased (Investigations) | 4 (8)
Anorexia (Metabolism and nutrition disorders) | 8 (10)
Dehydration (Metabolism and nutrition disorders) | 18 (31)
Hyperglycemia (Metabolism and nutrition disorders) | 7 (11)
Hyperkalemia (Metabolism and nutrition disorders) | 2 (3)
Hypernatremia (Metabolism and nutrition disorders) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 2 (2)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (1)
Hypoglycemia (Metabolism and nutrition disorders) | 2 (3)
Hypokalemia (Metabolism and nutrition disorders) | 1 (5)
Hypomagnesemia (Metabolism and nutrition disorders) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1)
Hypophosphatemia (Metabolism and nutrition disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 5 (6)
Musculoskeletal and connective tissue disorder - Other (Musculoskeletal and connective tissue disorders) | 3 (3)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2)
Neck pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Trismus (Musculoskeletal and connective tissue disorders) | 3 (4)
Akathisia (Nervous system disorders) | 1 (1)
Dizziness (Nervous system disorders) | 3 (3)
Dysgeusia (Nervous system disorders) | 42 (91)
Dysphasia (Nervous system disorders) | 1 (1)
Headache (Nervous system disorders) | 9 (11)
Myelitis (Nervous system disorders) | 2 (2)
Paresthesia (Nervous system disorders) | 1 (1)
Peripheral motor neuropathy (Nervous system disorders) | 1 (1)
Tremor (Nervous system disorders) | 1 (1)
Anxiety (Psychiatric disorders) | 2 (2)
Confusion (Psychiatric disorders) | 1 (2)
Depression (Psychiatric disorders) | 1 (1)
Hematuria (Renal and urinary disorders) | 1 (1)
Urinary frequency (Renal and urinary disorders) | 1 (1)
Urine discoloration (Renal and urinary disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Laryngeal hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Laryngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 5 (7)
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 8 (8)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1 (1)
Fat atrophy (Skin and subcutaneous tissue disorders) | 1 (1)
Nail loss (Skin and subcutaneous tissue disorders) | 2 (2)
Nail ridging (Skin and subcutaneous tissue disorders) | 3 (3)
Pain of skin (Skin and subcutaneous tissue disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 5 (5)
Rash acneiform (Skin and subcutaneous tissue disorders) | 35 (59)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1)
Scalp pain (Skin and subcutaneous tissue disorders) | 1 (1)
Skin and subcutaneous tissue disorders - Other (Skin and subcutaneous tissue disorders) | 2 (3)
Skin atrophy (Skin and subcutaneous tissue disorders) | 1 (1)
Skin ulceration (Skin and subcutaneous tissue disorders) | 1 (1)
Hypotension (Vascular disorders) | 1 (2)
Superficial thrombophlebitis (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-03-20): https://cdn.clinicaltrials.gov/large-docs/59/NCT01663259/Prot_SAP_000.pdf